CLINICAL TRIAL: NCT01594619
Title: An Open-label, Sequential, 3-period Study to Assess the Effects of Diltiazem on the Pharmacokinetics of Naloxegol in Healthy Subjects
Brief Title: Study in Healthy Volunteers to Investigate the Effects of Diltiazem on the Pharmacokinetics of Naloxegol
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: D3820C00032
Record Dates: First submitted 2012-05-08; First posted 2012-05-09 (Estimated); Last update posted 2014-10-15 (Estimated); Status verified 2014-10

CONDITIONS: Drug Induced Constipation
Keywords: Phase 1; Healthy male and female volunteers; Drug-drug interaction; Pharmacokinetics; Naloxegol
MeSH Terms: interventions — naloxegol; Diltiazem

ARMS (3):
- A (Experimental): Single dose naloxegol 25mg
  Interventions: Drug: Naloxegol
- B (Active Comparator): Diltiazem 240mg once daily day 4-6
  Interventions: Drug: Diltiazem XR
- C (Active Comparator): Diltiazem 240mg once daily day 7 and 8. Single dose naloxegol 25mg day 7
  Interventions: Drug: Naloxegol; Drug: Diltiazem XR

INTERVENTIONS:
Drug: Naloxegol — Oral 25mg tablet
  Arms: A; C
Drug: Diltiazem XR — Oral 240mg tablet
  Arms: B; C

SUMMARY:
Study in healthy volunteers to investigate the effects of Diltiazem on the Pharmacokinetics of naloxegol.

DETAILED DESCRIPTION:
An Open-label, sequential, 3-period study to Assess the Effects of Diltiazem on the Pharmacokinetics of Naloxegol in Healthy Subjects

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated, written informed consent prior to any study-specific procedures.
* Male and female (nonchildbearing potential, nonlactating) healthy volunteers aged 18 to 55 years inclusive, with suitable veins for cannulation or repeated venipuncture.
* Female volunteers must have negative pregnancy test (screening and admission), must not be lactating, and must be of nonchildbearing potential, confirmed at screening by being postmenopausal, or documentation of irreversible surgical sterilization not in.
* Male volunteers should be willing to use barrier contraception ie, condoms, from the first day of dosing until 3 months after dosing with the IP. The female partner should use contraception during this period.
* Volunteers must have a BMI between 18 and 30 kg/m2, inclusive, and weigh at least 50 kg.

Exclusion Criteria:

* Any clinically significant disease or disorder (eg, cardiovascular, pulmonary, gastrointestinal, liver, renal, neurological, musculoskeletal, endocrine) which, may put the volunteer at risk of participation in the study, or influence of the ADME of drugs.
* Any clinically significant illness, medical/surgical procedure or trauma within 4 weeks of the first administration of IP.
* Any clinically significant abnormalities in clinical chemistry, hematology, or urinalysis results as judged by the Investigator.
* Significant orthostatic reaction at enrolment, as judged by the Investigator.
* Abnormal vital signs, after 10 minutes supine rest as defined in protocol.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2012-05; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Description of the pharmacokinetic (PK) profile for naloxegol in terms of maximum observed plasma concentration (Cmax) and area under the plasma concentration-time curve from time zero extrapolated to infinity (AUC). | At predose on Days 1 and 7 and then at 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 16, 24, 36, 48, and 72 hours postdose

SECONDARY OUTCOMES:
Description of the safety profile in terms of adverse events, clinical laboratory assessments , vital signs (blood pressure and pulse rate), physical examinations, electrocardiograms, and Columbia-Suicide Severity Rating scale | From baseline day 1 through to Follow-up (Maximum 21 days)
Description of the pharmacokinetic (PK) profile for naloxegol in terms of time to Cmax (tmax), terminal half-life (t1/2λz), terminal rate constant (λz). | At predose on Day 1 and 7 and then at 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 16, 24, 36, 48, and 72 hours postdose
Description of the pharmacokinetic (PK) profile for naloxegol in terms of area under the plasma concentration-time curve from time zero to the time of the last quantifiable concentration [AUC(0-t)]. | At predose on Day 1 and 7 and then at 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 16, 24, 36, 48, and 72 hours postdose
Description of the pharmacokinetic (PK) profile for naloxegol in terms of area under the plasma concentration-time curve from time zero to 24hours postdose [AUC(0 24)]. | At predose on Day 1 and 7 and then at 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 16, 24, 36, 48, and 72 hours postdose
Description of the pharmacokinetic (PK) profile for naloxegol in terms of apparent oral clearance from plasma (CL/F), and apparent volume of distribution during the terminal phase (Vz/F) | At predose on Day 1 and 7 and then at 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 16, 24, 36, 48, and 72 hours postdose

CONTACTS AND LOCATIONS:
Overall Officials: Bo Fransson, MD, Study Chair — AstraZeneca, Sodertalje Sweden; Dave Matthews, MD, Principal Investigator — Quintiles, Inc Kansas Overland Park US; Mark Sostek, MD, Study Director — AstraZeneca, Wilmington US
Locations (1):
- Research Site, Overland Park, Kansas, United States

REFERENCES:
- See also: Clinical_Study_Report_Synopsis_D3820C00032 — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=1401&filename=Clinical_Study_Report_Synopsis_D3820C00032.pdf